CLINICAL TRIAL: NCT07283900
Title: Title: A Phase II Trial of High Dose Ascorbate in Combination With Azacitidine in Adults With Myelodysplastic Syndrome
Brief Title: Ascorbate in Myelodysplastic Syndrome
Acronym: AIMS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prajwal Dhakal (Other)
Responsible Party: Sponsor-Investigator, Prajwal Dhakal, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202508099
Record Dates: First submitted 2025-11-19; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: Vitamin C; Ascorbate; Myelodysplastic Syndrome; AIMS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Ascorbic Acid; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- High-Dose Ascorbate + Azacitidine (Experimental): All participants receive the combination of high-dose intravenous ascorbate (75 g on days 1, 3, 5, and 7) and azacitidine (75 mg/m² intravenous or subcutaneous on days 1-7) in 28-day treatment cycles.
  Interventions: Drug: High-dose ascorbate; Drug: Azacitidine

INTERVENTIONS:
Drug: High-dose ascorbate — Ascorbate, or vitamin C, is a water-soluble vitamin with antioxidant properties that also functions as a cofactor for several enzymatic reactions, including collagen synthesis and the activity of dioxygenase enzymes involved in DNA and histone demethylation
  Other Names: Vitamin C
Drug: Azacitidine — Azacitidine is a pyrimidine nucleoside analog of cytidine that incorporates into RNA and DNA, inhibiting DNA methyltransferase and leading to global DNA hypomethylation
  Other Names: Vidaza

SUMMARY:
This is an open-label, phase II clinical trial with safety run-in evaluating the safety, tolerability, and efficacy of IV HDA in combination with azacitidine for participants with MDS.

DETAILED DESCRIPTION:
This Phase II clinical trial investigates the combination of high-dose intravenous ascorbate (vitamin C) with azacitidine in adults with higher-risk myelodysplastic syndrome (MDS). The study includes a small safety run-in followed by an efficacy phase, enrolling a total of 38 participants. It aims to determine whether adding high-dose ascorbate can safely enhance the therapeutic response to azacitidine, a standard hypomethylating agent used in MDS treatment.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Diagnosis of myelodysplastic syndrome (MDS) requiring treatment with a hypomethylating agent (HMA).
* Higher-risk MDS per the Molecular International Prognostic Scoring System (IPSS-M) - Moderate High, High, or Very High risk categories.
* No prior MDS-directed therapy, except:

  ≤ 1 prior cycle of azacitidine, decitabine, or oral decitabine-cedazuridine; or prior use of ESA, luspatercept, or imetelstat. Prior hydroxyurea use is allowed but continuation beyond Cycle 1 requires PI approval.
* ECOG performance status 0-2.
* Adequate organ function: Creatinine clearance >45 mL/min; total bilirubin ≤1.5 × ULN; ALT and AST ≤3 × ULN.
* Ability to provide written informed consent.
* Willingness to comply with study visits, treatment, and contraception requirements.
* Negative pregnancy test for women of childbearing potential at screening.

Exclusion Criteria

* MDS with isolated del(5q) eligible for lenalidomide therapy.
* MDS/MPN overlap syndromes other than MDS.
* Known hypersensitivity or allergy to ascorbate or azacitidine.
* Pregnant or nursing individuals.
* Inability or unwillingness to use adequate contraception.
* Uncontrolled intercurrent illness including active infection, recent myocardial infarction (≤6 months), uncontrolled heart failure or arrhythmia, pulmonary edema, unstable angina, or significant psychiatric illness.
* Renal disease requiring dialysis, diabetic nephropathy, renal transplant recipients, or history of oxalate nephropathy.
* Paroxysmal nocturnal hemoglobinuria.
* Uncontrolled HIV infection (patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible).
* G6PD deficiency.
* Use of warfarin (due to potential interaction with high-dose ascorbate).
* Diabetic patients using fingerstick or continuous glucose monitors to adjust insulin doses (ascorbate can cause false readings).
* Concurrent active malignancy, except adequately treated nonmelanoma skin cancer or curatively treated in situ cancers with >2 years disease-free.
* Systemic immunosuppressive therapy with prednisone ≥20 mg/day (or equivalent), except for inhaled or topical steroids.
* Primary hemochromatosis or transfusion-related iron overload (ferritin >1000 ng/mL).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | At the end of Cycle 1 (each cycle is 28 days)
  Assess the safety and tolerability of intravenous (IV) high-dose ascorbate (HDA) in combination with azacitidine.
Treatment Efficacy | At the end of Cycle 4 (each cycle is 28 days)
  Proportion of participants achieving a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Overall Survival (OS) | From treatment initiation until death from any cause or up to 24 months, whichever comes first
  Time from treatment initiation to death from any cause.
Event-Free Survival (EFS) | From treatment initiation until disease progression, disease relapse, treatment failure, or death from any cause, whichever came first, assessed up to 24 months
  Time from treatment initiation to progression, relapse, treatment failure, or death.
Transfusion Requirements | At baseline, assessed throughout the treatment up to the end of cycle 4 (each cycle is 28 days)
  Changes in red blood cell and platelet transfusion needs during treatment.
Hematologic Parameters | At baseline, assessed throughout the treatment up to the end of cycle 4 (each cycle is 28 days)
  Changes in hemoglobin, platelet, and neutrophil counts.
Composite Complete Response (cCR) Rate | At the end of cycle 4 (each cycle is 28 days)
  Proportion of participants achieving CR, CRh, CRL, or CR-equivalent per IWG 2023 criteria.
Overall Response Rate (ORR) | At the end of cycle 4 (each cycle is 28 days)
  Proportion of participants achieving CR, CRh, CRL, PR, or hematologic improvement (HI) per IWG 2023 criteria after four treatment cycles
Health-Related Quality of Life (HRQOL) Using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | At baseline, at the end of cycle 4, every 3 months after the end of cycle 4 up to 24 months (each cycle is 28 days)
  HRQOL will be assessed using the EORTC QLQ-C30 questionnaire. This outcome measure will evaluate participants' overall quality of life, functional status, and symptom burden at various time points throughout the study. Scoring Range: 0 to 100 for each scale. Functioning Scales: Higher scores = better functioning. Symptom Scales: Higher scores = worse symptoms. Global Health Status/QOL Scale: Higher scores = better overall QOL.
Health-Related Quality of Life (HRQOL) using EuroQol (EQ-5D-5L) questionnaire | At baseline, at the end of cycle 4, every 3 month after end of cycle 4 up to 24 months (each cycle is 28 days)
  HRQOL will be assessed using the EQ-5D-5L questionnaire, which uses a descriptive system and a visual analogue scale. The descriptive system will evaluate participants' mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scoring range: 11111 to 55555. Higher scores= worse problems. The visual analog scale asks patients to rate their current health on a scale of 0 to 100. Higher scores= better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Prajwal Dhakal, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States